CLINICAL TRIAL: NCT03635073
Title: A Phase 2, Prospective, Interventional, Open-Label, Multi-Site, Extension Study to Assess the Long-Term Safety and Tolerability of Soticlestat (TAK-935) as Adjunctive Therapy in Subjects With Developmental Epileptic Encephalopathies Including Dravet Syndrome, Lennox Gastaut Syndrome, CDKL5 Deficiency Disorder, and Chromosome 15 Duplication Syndrome (ENDYMION 1)
Brief Title: A Study of Soticlestat in Adults and Children With Rare Epilepsies
Acronym: Endymion 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to negative results from phase 3 SKYLINE and SKYWAY studies and unrelated to patient safety it has been determined that supplementary data from TAK-935-18-001 study is no longer necessary. Therefore, Takeda has made a decision to close this study
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-935-18-001; U1111-1218-5515 (Other: WHO); 2018-002485-39 (EudraCT Number); 2022-502801-13-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2018-08-06; First posted 2018-08-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Dravet Syndrome (DS); Lennox-Gastaut Syndrome (LGS)
Keywords: Soticlestat; Drug Therapy
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Soticlestat (Experimental): Treatment: Soticlestat, tablets orally twice daily at optimized dose, titrated in up to 2 weeks of Dose Optimization Period, followed by Maintenance Period, which lasts until development is stopped by the sponsor, or the product is approved for marketing, or at any time at the discretion of the sponsor.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets or mini-tablets.
  Other Names: TAK-935

SUMMARY:
The main aim is to assess the long-term safety and tolerability of soticlestat when used along with other anti-seizure treatment.

Participants will receive soticlestat twice a day. Participants will visit the study clinic every 2-6 months throughout the study.

Study treatments may continue as long as the participant is receiving benefit from it.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). This global, open-label extension (OLE) study will assess the long-term safety and tolerability of soticlestat in participants with developmental and epileptic encephalopathy (DEE) who participated in previous short-term efficacy/safety studies of soticlestat. All participants will receive Soticlestat treatment.

Participants who rollover from previous blinded study will undergo up to 2 weeks of Dose Optimization Period (depending on the previous study) followed by Maintenance Period. Participants who rollover from an open-label study will continue on their current dose until development is stopped by the sponsor, or the product is approved for marketing, or at any time at the discretion of the sponsor. There will be a 4-week Safety Follow-up Period after the last dose in Maintenance Period, including a 2-week dose Tapering Period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have participated in a previous soticlestat study and meet one of the following conditions:

   * Successfully completed a soticlestat clinical study.
   * Received at least 10 weeks of treatment with the study drug in an antecedent placebo-controlled blinded soticlestat clinical study and the participant did not have a serious or severe AE that, in the investigator's or sponsor's opinion, was related to the study drug and would make it unsafe for the participant to continue receiving the study drug.
2. In the opinion of the investigator, the participant has the potential to benefit from the administration of soticlestat

Exclusion Criteria:

1. Clinically significant disease, that, in the investigator's opinion, precludes study participation.
2. Enrollment in any other clinical trial involving an investigational drug, device, or treatment in the past 90 days (with the exception of an antecedent study involving Soticlestat).
3. Participant is currently pregnant or breastfeeding or is planning to become pregnant during the study or within 30 days of the last study drug administration.
4. Suicide attempt within the last year, at significant risk of suicide (either in the opinion of the investigator or defined as 'yes' to suicidal ideation question 4 or 5 on the C-SSRS at Screening) or appearing suicidal per investigator judgment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience At least one Adverse Event (AE) | Up to 6 years
  An Adverse Event (AE) is defined any untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable or unintended sign (for example, an abnormal laboratory finding, vital sign or ECG evaluation), symptom, or disease temporally associated with the use of a medicinal product, whether considered related to this medicinal product.
Change from Baseline in Behavioral and Adaptive Functional Measures Using the Vineland Adaptive Behavior Scale (VABS) | Up to 6 years
  The VABS, 3rd edition, Parent Caregiver Form (VABS-3 Parent Caregiver Form), is a parent-report questionnaire of adaptive functioning or how an individual behaves in their day-to-day life at home and in the community.
Change from Baseline in Behavior Measures Using Total Scores and Subscale Scores of the Aberrant Behavior Checklist-Community Edition (ABC-C) for Participants ≥6 Years of age | Up to 6 years
Change from Baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) Categorization Based on Columbia Classification Algorithm of Suicide Assessment Categories 1,2,3,4, and 5 for Participants ≥6 Years of age | Up to 6 years

SECONDARY OUTCOMES:
Percent Change from Baseline in all Seizure 28-day Frequency | Up to 6 years
Percent Change from Baseline in Drop Seizure 28-day Frequency (Lennox-Gastaut syndrome [LGS] Participants) | Up to 6 years
Percent Change from Baseline in Convulsive Seizure 28-day Frequency (Dravet syndrome [DS] Participants) | Up to 6 years
Percent Change from Baseline in Motor Seizure 28-day Frequency | Up to 6 years
Change from Baseline in Clinician's Clinical Global Impression of Severity (CGI-S) | Up to 6 years
  CGI-S is used to obtain an assessment of symptom severity, focusing on clinicians' observations of the subject's current cognitive, functional, and behavioral performance. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill participants).

CONTACTS AND LOCATIONS:
Locations (51):
- United States (22):
  - Xenosciences Inc, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Pediatric Neurology PA, Winter Park, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Bluegrass Epilepsy Research LLC, Lexington, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic - PIN, Rochester, Minnesota
  - Minnesota Epilepsy Group PA, Saint Paul, Minnesota
  - Max Benzaquen, M.D., PC, Chesterfield, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Children's Hospital at Saint Peter's University Hospital, New Brunswick, New Jersey
  - NYU - Ambulatory Care Center (ACC), New York, New York
  - Columbia University Medical Center - PIN, New York, New York
  - Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - Medical University of South Carolina Childrens Hospital - PIN, Charleston, South Carolina
  - Cook Children's Medical Center - Jane and John Justin Neurosciences Center, Fort Worth, Texas
- Australia (3):
  - Monash Children's Hospital, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Austin Hospital, Heidelberg West, Victoria
- Hospital For Sick Children, Toronto, Ontario, Canada
- China (6):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Peking University First Hospital, Beijing
  - Beijing Children's Hospital,Capital Medical University, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
- Israel (7):
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv, Tel Aviv
  - Soroka University Medical Centre, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Schneider Children's Medical Center of Israel - Petah Tikvah - PIN, Petah Tikva
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Poland (5):
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Plejady, Krakow
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny w Warszawie, Warsaw
  - NZOZ Centrum Neurologii Dzieciecej i Leczenia Padaczki, Kielce, Świętokrzyskie Voivodeship
- Portugal (2):
  - Centro Hospitalar Lisboa Central- Hospital Dona Estefania, Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. Hospital de Santa Maria, Lisbon
- Spain (5):
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid, Madrid, Communidad Delaware
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Vithas La Salud, Granada
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/517cf1e47a6a477f?idFilter=%5B%22TAK-935-18-001%22%5D